CLINICAL TRIAL: NCT03804840
Title: A Mobile Prototype for a Field Sobriety Test for Cannabis
Brief Title: Developing a Mobile Method to Measure THC-induced Impairment
Acronym: AIS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB16-1132a
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Measuring THC-induced Cognitive Impairment Using a Mobile Application
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 7.5 mg THC (Active Comparator)
  Interventions: Drug: Dronabinol
- 15 mg THC (Active Comparator)
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — THC (Marinol® [dronabinol]; Solvay Pharmaceuticals) will be orally administered in doses of 7.5 mg and 15 mg, in opaque capsules with dextrose filler. Placebo capsules contain only dextrose. These doses of THC are known to produce performance impairments as well as subjective intoxication.
  Arms: 15 mg THC; 7.5 mg THC
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Marijuana use, for both recreational and therapeutic purposes, is becoming increasingly common as states remove restrictions on use. The increased use raises new concern about the safety of this drug, including its ability to impair basic cognitive and psychomotor tasks, and whether the users are aware of their impairment. We propose to design a simple performance test that users can use in the field, using a cell phone, to assess their level of impairment relative to their own drug-free state. In this preliminary study, we will compare participants' simple task performance after a known dose of delta-9-tetrahydrocannabinol (THC), or placebo, administered under double-blind conditions. In our app the participants will be asked to gauge their own perceived level of impairment (as determined by self-ratings and judgments of impairment) as well as their actual impairment (as gauged by the app), providing important feedback and training about their ability to detect impairment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-35 years old, males and females (N=44; 36 completers; 18 men, 18 women)
2. BMI 19-26
3. High school education, fluent in English
4. Experienced non-daily marijuana users

   Exclusion Criteria:
5. Current drug/alcohol abuse or dependence
6. Past year drug/alcohol dependence
7. Diagnosis with drug treatment for psychosis/bipolar/schizophrenia
8. Past year major depression
9. Panic/anxiety attacks in past 2 months
10. Post Traumatic Stress Disorder
11. Attention Deficit Hyperactivity Disorder
12. Cardiovascular illness, high blood pressure, abnormal EKG
13. Current medications
14. Pregnant or planning to become pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Pabon, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Broyd SJ, van Hell HH, Beale C, Yucel M, Solowij N. Acute and Chronic Effects of Cannabinoids on Human Cognition-A Systematic Review. Biol Psychiatry. 2016 Apr 1;79(7):557-67. doi: 10.1016/j.biopsych.2015.12.002. Epub 2015 Dec 8. PMID 26858214
- [Result] Hartman RL, Huestis MA. Cannabis effects on driving skills. Clin Chem. 2013 Mar;59(3):478-92. doi: 10.1373/clinchem.2012.194381. Epub 2012 Dec 7. PMID 23220273

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
Started | 24 | 24 | 24
Completed | 24 | 24 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 7.5 mg THC; 15 mg THC: Dronabinol: THC (Marinol® [dronabinol]; Solvay Pharmaceuticals) will be orally administered in doses of 7.5 mg and 15 mg, in opaque capsules with dextrose filler. Placebo capsules contain only dextrose. These doses of THC are known to produce performance impairments as well as subjective intoxication (Broyd et al, 2016; Hartman and Huestis, 2013).
- Total: Total of all reporting groups
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 24 | 72
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 12 | 36
  Male | 12 | 12 | 12 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 12
  White | 12 | 12 | 12 | 36
  More than one race | 4 | 4 | 4 | 12
  Unknown or Not Reported | 2 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 24 | 72
Education - High School Education [Count of Participants; unit: Participants] | 24 | 24 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Simple Reaction Time
Description: In this reaction time task, the user is asked to shake the device in response to a visual clue on the device's screen. The user makes three attempts, in which he or she must shake or move the device with an acceleration that is greater than the value of the thresholdAcceleration property within the given time. The task finishes when the user successfully completes the attempts as instructed in the task. Data collected by this task is in the form of ORKReactionTimeResult objects. Each of these objects contain a timestamp representing the delivery of the stimulus and an ORKFileResult object that references the motion data collected during an attempt.
Time Frame: Assessed two hour post intervention at peak effects
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
Number analyzed (Participants) | 24 | 24 | 24
Seconds | .365 (.07) | .386 (.09) | .396 (.10)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 weeks
Arm/Group | Placebo | 7.5 mg THC | 15 mg THC
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03804840/Prot_SAP_000.pdf